CLINICAL TRIAL: NCT01436357
Title: A Staged Phase I/II Study, to Assess Safety, Efficacy and Immunogenicity of a New Hepatitis C Prophylactic Vaccine Based on Sequential Use of AdCh3NSmut1 and MVA-NSmut
Brief Title: Staged Phase I/II Hepatitis C Prophylactic Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10-0069
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2017-04-05

CONDITIONS: Hepatitis C
Keywords: AdCh3NSmut1; Hepatitis C; MVA-NSmut; vaccine
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Stage I and II) (Experimental): Receive AdCh3NSmut1 at 2.5 x 10^10 total virus particles (vp)/dose at day 0 followed by 1 dose of MVA-NSmut intramuscularly 56 days later at the dosage 1.8 x10^8 plaque forming units (pfu): 34 (+/-2) subjects Stage I, then 191 (+/-2) subjects at Stage II.
  Interventions: Biological: AdCh3NSmut1; Biological: MVA-NSmut
- Arm B (Stage I and II) (Placebo Comparator): Two doses of placebo intramuscularly, 1 at day 0 and 1 at day 56: 34 (+/-2) subjects Stage I, then 191 (+/-2) subjects at Stage II.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AdCh3NSmut1 — Stages I and II: Receive AdCh3NSmut1 at 2.5 x 10^10 total virus particles (vp)/dose, intramuscularly on day 0.
  Arms: Arm A (Stage I and II)
Biological: MVA-NSmut — Stages I and II: 1 dose of MVA-NSmut at the dosage 1.8 x10^8 plaque forming units (pfu) intramuscularly on day 56.
  Arms: Arm A (Stage I and II)
Other: Placebo — Stages I and II: Two doses of placebo intramuscularly, 1 at day 0 and 1 at day 56.
  Arms: Arm B (Stage I and II)

SUMMARY:
A two stage, phase I/II, double-blinded, randomized, placebo-controlled study of hepatitis C virus (HCV)uninfected male and female injection drug users (IDU) aged 18 to 45. AdCh3NSmut1 and MVA-NSMut HCV vaccine will be administered to 68 (+/-4) volunteers in stage 1. A planned interim analysis of safety and immunogenicity will be conducted. If no safety signal is detected and there is evidence of a measurable immune response to HCV then 472 (+/-4) volunteers will be enrolled in stage 2. Primary objectives are to 1) assess the safety of AdCh3NSmut1 and MVA-NSmut compared to placebo when administered to HCV-uninfected IDUs and 2) determine if AdCh3NSmut1 and MVA-NSmut HCV vaccines will reduce incidence of chronic HCV infection compared to placebo among HCV-uninfected IDUs. Planned study duration is approx 63 months (accrual time, 2 months vaccination, 18 months follow-up, and 9 months extended observation for subjects becoming viremic in the last month of follow-up).

DETAILED DESCRIPTION:
A two stage, phase I/II, double-blinded, randomized, placebo-controlled study of hepatitis C virus (HCV)uninfected male and female injection drug users (IDU) aged 18 to 45. In this clinical trial AdCh3NSmut1 and MVA-NSMut HCV vaccine will be administered intramuscularly to 68 (+/-4) evaluable volunteers in stage 1. A planned interim analysis of safety and immunogenicity will be conducted based on data through 1 week after receipt of the second vaccination. If no safety signal is detected and there is evidence of a measurable immune response to HCV then an additional 472 (+/-4) volunteers will be enrolled in stage 2. The primary objectives of this study will be 1) to assess the safety of the new candidate hepatitis C virus vaccines, AdCh3NSmut1 and MVA-NSmut, compared to placebo when administered to HCV-uninfected injection drug users (IDUs) and 2) to determine if AdCh3NSmut1 and MVA-NSmut HCV vaccines will reduce incidence of chronic HCV infection compared to placebo among HCV-uninfected IDUs. The secondary objective of this study will be to evaluate the immunogenicity of the new candidate hepatitis C virus vaccines, AdCh3NSmut1 and MVA-NSmut, compared to placebo when administered to HCV-uninfected IDUs.The planned duration of the study is approximately 63 months total including accrual time for subjects (assuming 31 months of screening/enrollments, plus 3 months of halted enrollment for the first interim analysis), 2 months vaccination, 18 months follow-up of each enrolled subject, and 9 months extended observation (monthly), from the time of infection, for subjects becoming viremic in the last month of follow-up.

ELIGIBILITY:
Inclusion Criteria:

- Comprehension of informed consent. - 18-45 year old men or women with acknowledged active IDU in the past 90 days and have no travel plans that would interfere with ability to meet the study visit schedule. - In good general health as determined by a participating study physician and results within acceptable ranges for clinical laboratory evaluations as detailed in Appendix A. - Negative for antibodies to hepatitis C virus (anti-HCV). - Negative for HCV RNA. - Negative antibodies to HIV. - Negative for HBsAg. - Able and willing (in the Investigator's opinion) to comply with all study requirements. - Willing to allow the investigators access to their medical records. - Willingness to practice continuous effective contraception from the screening visit through 90 days after the last vaccination (males and females). - Among females, a negative pregnancy test within 24 hours prior to vaccination. - Agreement to refrain from blood donation during the course of the study or after the study. - Provide written informed consent prior to initiation of any study procedures. - Willing to provide contact information for study follow-up activities, including the address, name and contact information of three people who can be contacted to facilitate follow-up compliance.

Exclusion Criteria:

- The subject is currently participating in a study that involves an experimental agent (vaccine, drug, biologic device, blood product, or medication) or has received an experimental agent within 30 days prior to enrollment in this study, or expects to receive another experimental agent during participation in this study. - Prior receipt of a recombinant simian or human adenoviral vaccine or MVA vaccine. - Administration of immunoglobulins and/or any blood products within the 90 days preceding the planned administration of the vaccine candidate. - Any confirmed or suspected immunosuppressive or immunodeficient state, including: HIV infection; asplenia; recurrent, severe infections. - History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (i.e., known hypersensitivity to aminoglycosideantibiotics or to egg proteins). - History of clinically significant contact dermatitis or other significant dermatological conditions such as psoriasis. - Any history of anaphylaxis in reaction to vaccination. - Pregnancy, lactation or willingness/intention to become pregnant during the study. - History of cancer (except for successfully treated basal cell carcinoma of the skin and cervical carcinoma in situ). - History of severe psychiatric illness, including severe depression, history of suicidal ideation, suicidal attempts, or psychosis requiring medication. The subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis that is uncontrolled and would interfere with the ability to adhere to the protocol. - Any other serious chronic illness requiring hospital specialist supervision. - Suspected or known current alcohol abuse as defined by a score of 10 or more on the Alcohol Use Disorders Identification Test (AUDIT) C test (a standardized screening tool used to identify hazardous drinkers or those with active alcohol use disorders, including abuse or dependence). - At high risk of HIV infection by the following criteria (adapted from HIV Network for Prevention Trials (HIVNET) behavioral criteria for high risk of HIV): (1) sexually active male who has sex with men (MSM), defined as (i) male who has had anal sex with male sexual partner or partners in the past year or (ii) a male who exchanged sex with male partner(s) for money or drugs in the past year; and (2) female and in a current relationship with a high risk male (active MSM, HIV positive male). - Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, may influence the result of the study, or may influence the subject's ability to participate in the study. - History of or current diagnosis of Diabetes mellitus. - History of or current diagnosis of autoimmune disease. - History of or current cardiac disease including history of myocardial infarction or arrhythmia. - Current diagnosis of active liver disease. - History of seizure disorder or currently taking anti-convulsant therapy that would interfere with safety evaluation. - Uncontrolled hypertension (defined as systolic blood pressure being greater than 140mm Hg or diastolic blood pressure being greater than 90mm Hg). - History of splenectomy. - Long term immunosuppressive use (defined as taken for 14 days or more in total at any time during the past 180 days) of high dose oral or parenteral glucocorticoids (high dose defined as prednisone >/=20 mg total daily dose, or equivalent dose of other glucocorticoids); or high-dose inhaled steroids (high dose defined as >800 mcg/day of beclomethasone dipropionate or equ ivalent); or any use of hepatotoxic or non-FDA approved medication. - Have an acute illness, including an oral temperature greater than or equal to 100.4 degrees Fahrenheit, within 7 days prior to the first vaccination. - Immunization against another pathogen within 14 days of planned injection. Second vaccination exclusion criteria: The following events associated with vaccine immunization constitute absolute contraindications to further administration of vaccine. The subject will not receive additional vaccination, but will continue with scheduled follow-up procedures except vaccination. 1. Anaphylactic reaction following administration of vaccine. 2. Pregnancy. If a woman reports having a positive home urine pregnancy test or a positive in clinic urine pregnancy test prior to a scheduled second vaccination, she is not eligible to receive the study vaccine. If she later returns to clinic and reports having a negative home urine pregnancy test and this is confirmed by a negative in clinic urine pregnancy test and a negative blood pregnancy test she may be eligible for the second vaccination if she is still within the vaccination window and no other exclusion criteria are met. The following adverse events constitute contraindications to administration of vaccine at that point in time. If any one of these adverse events occurs at the time scheduled for vaccination, the subject may be vaccinated at a later date (within 28 days of scheduled administration) or withdrawn at the discretion of the investigator. The subject will not receive additional vaccination, but will continue with all scheduled follow-up procedures except vaccination. 3. Acute disease at the time of vaccination (acute disease is defined as the presence of a moderate or severe illness with or without fever). The vaccine dose can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., temperature of <38°C (100.4°F). 4. Temperature of >38°C (100.4°F) at the time of vaccination. 5. Immunization against another pathogen within 14 days of vaccination

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 548 (Actual)
Dates: Start 2012-03-06 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California San Francisco - Tenderloin Clinical Research Center, San Francisco, California
  - UCSF Community Research Center, San Francisco, California
  - Zuckerberg San Francisco General Hospital Unit 5B, San Francisco, California
  - Johns Hopkins School of Public Health - Wood Clinic, Baltimore, Maryland
  - University of New Mexico - Truman Health Services, Albuquerque, New Mexico

REFERENCES:
- [Derived] Page K, Melia MT, Veenhuis RT, Winter M, Rousseau KE, Massaccesi G, Osburn WO, Forman M, Thomas E, Thornton K, Wagner K, Vassilev V, Lin L, Lum PJ, Giudice LC, Stein E, Asher A, Chang S, Gorman R, Ghany MG, Liang TJ, Wierzbicki MR, Scarselli E, Nicosia A, Folgori A, Capone S, Cox AL. Randomized Trial of a Vaccine Regimen to Prevent Chronic HCV Infection. N Engl J Med. 2021 Feb 11;384(6):541-549. doi: 10.1056/NEJMoa2023345. PMID 33567193
- [Derived] Salinas E, Boisvert M, Upadhyay AA, Bedard N, Nelson SA, Bruneau J, Derdeyn CA, Marcotrigiano J, Evans MJ, Bosinger SE, Shoukry NH, Grakoui A. Early T follicular helper cell activity accelerates hepatitis C virus-specific B cell expansion. J Clin Invest. 2021 Jan 19;131(2):e140590. doi: 10.1172/JCI140590. PMID 33463551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: People who are actively injecting drugs who are at high risk for HCV infection, negative for HCV antibodies and HCV RNA at screening, were recruited at 3 clinical sites experienced in recruiting and retaining people who inject drugs in prospective studies. Participants were enrolled between 19MAR2012 and 28OCT2016.
Groups:
- AdCh3NSmut1 and MVA-NSmut: One dose of AdCh3NSmut1 at 2.5 x 10^10 total virus particles (vp)/dose at day 0 followed by 1 dose of MVA-NSmut intramuscularly 56 days later at the dosage 1.8 x10^8 plaque forming units (pfu).
- Sodium Chloride Placebo: Two doses of sodium chloride placebo intramuscularly, 1 at day 0 and 1 at day 56.
Period: Overall Study
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Started | 274 | 274
Stage 1 | 49 | 48
Stage 2 | 225 | 226
Completed | 152 | 146
Not Completed | 122 | 128
Not completed — Death | 5 | 1
Not completed — Enrolled but not vaccinated | 1 | 1
Not completed — Incarceration | 18 | 20
Not completed — Lost to Follow-up | 67 | 61
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 26 | 38
Not completed — Physician Decision | 3 | 4
Not completed — Moved out of area | 1 | 2
Not completed — Subject in rehab | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo | Total
Number analyzed (Participants) | 274 | 274 | 548
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 274 | 274 | 548
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (7.3) | 30.4 (7.2) | 30.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 214 | 212 | 426
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 39 | 79
  Not Hispanic or Latino | 234 | 235 | 469
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 2 | 9
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 62 | 51 | 113
  White | 159 | 175 | 334
  More than one race | 33 | 30 | 63
  Unknown or Not Reported | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 274 | 274 | 548
IL28B Status [Count of Participants; unit: Participants] — The IL28B gene is involved in the immune response to certain viruses, including hepatitis C. There are three IL28B subtypes (called genotypes): CC, CT, and TT. People with the CC genotype have a more potent immune response to HCV infection than people with the CT or TT genotypes (called non-CC genotypes). This immune response makes people who have a CC genotype more likely to clear HCV without treatment (called spontaneous viral clearance), within months of becoming infected. Given the impact of this gene, subjects were stratified based on having CC on non-CC genotypes.
  Participants
    CC | 111 | 111 | 222
    CT/TT | 163 | 163 | 326

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Chronic Hepatitis C Virus (HCV) Infection at 6 Months
Description: Chronic hepatitis C virus (HCV) infection was defined by persistent viremia over a period of 6 months after initial detection of primary infection.
Time Frame: 6 months
Population: All randomized are included as treated (one participant randomized to placebo received vaccine) with the following censoring criteria applied: did not receive both vaccinations, HCV infected at baseline, did not have sufficient follow-up to be evaluable for efficacy, or had major protocol deviations compromising the assessment of vaccine efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 275 | 273
Participants | 14 | 14
Statistical Analysis 1: Comparison: AdCh3NSmut1 and MVA-NSmut vs Sodium Chloride Placebo; Test type: Superiority; p = 0.317, Regression, Cox; Hazard Ratio (HR) = 1.529, 95% CI 2-sided [0.661 to 3.535]

2. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events (AEs) at 1 Month After First Vaccination
Description: Blood was collected at baseline and 1 month after each vaccination for assessment of alanine transferase (ALT) (SGPT), creatinine, hemoglobin, platelets, and white blood cells (WBC). A laboratory AE was defined for ALT as greater than 1.25 times the upper limit of normal. A laboratory AE was defined for creatinine as greater than or equal to 1.2 times the upper limit of normal (as appropriate for age and sex). A laboratory AE was defined for hemoglobin as less that or equal to 12.4 g/dl for males and less than or equal to 10.8 g/dl for females. A laboratory AE was defined for platelets as less than or equal to 117,000 per cumm. A laboratory AE was defined for WBC as less than or equal to 2.9 thou/mcl or greater than or equal to 11.9 thou/mcl.
Time Frame: 1 month after first vaccination
Population: The safety analysis population includes all participants with blood collected at the timepoint summarized. Participants are analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 274 | 272
Participants | 70 | 48
Statistical Analysis 1: Comparison: AdCh3NSmut1 and MVA-NSmut vs Sodium Chloride Placebo; Test type: Superiority; p = 0.029, Fisher Exact; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.01 to 0.16]

3. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events (AEs) at 1 Month After Second Vaccination
Description: as for outcome 2
Time Frame: 1 month after second vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 228 | 227
Participants | 73 | 49
Statistical Analysis 1: Comparison: AdCh3NSmut1 and MVA-NSmut vs Sodium Chloride Placebo; Test type: Superiority; p = 0.015, Fisher Exact; Risk Difference (RD) = 0.10, 95% CI 2-sided [0.01 to 0.20]

4. Primary Outcome: Number of Participants With Severe Local and/or Systemic Solicited Reactogenicity Signs and Symptoms in the 8 Days (Day 0-7) After First Vaccination
Description: Participants recorded temperature and the presence and intensity of post-vaccination reactogenicity events daily on an 8-day memory aid. Local solicited reactogenicity events included pain, tenderness, erythema, induration and warmth at the injection site. Systemic solicited reactogenicity events included fever, chills, arthralgia/joint pain, malaise/fatigue, myalgia/body aches, headache, nausea, vomiting, abdominal pain. Severe was defined as "events interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating." Measured erythema and induration of >50 mm and oral temperature >40.0 degrees Celsius were considered severe.
Time Frame: 7 days after first vaccination
Population: The safety analysis population includes all participants receiving the vaccination for whom data were available. Participants are analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 274 | 272
Participants | 0 | 0
Statistical Analysis 1: Comparison: AdCh3NSmut1 and MVA-NSmut vs Sodium Chloride Placebo; Test type: Superiority; p = 0.00, Fisher Exact; Risk Difference (RD) = 0.0

5. Primary Outcome: Occurrence of Vaccine-related Serious Adverse Events (SAEs) From the Time of First Vaccination Through the Entire Study Period
Description: The occurrence of SAEs was assessed at every study visit. The occurrence of SAEs may also have come to the attention of the investigator by secondary contacts of the participant when they did not present for study visits. Relationship to vaccine was assessed by the site investigator.
Time Frame: Day 0 to 29 months
Population: The safety analysis population excludes 1 participant who was not vaccinated. Participants are analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 274 | 272
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Severe Local and/or Systemic Solicited Reactogenicity Signs and Symptoms in the 8 Days (Day 0-7) After Second Vaccination
Description: as for outcome 4
Time Frame: 7 days after second vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 228 | 227
Participants | 2 | 0
Statistical Analysis 1: Comparison: AdCh3NSmut1 and MVA-NSmut vs Sodium Chloride Placebo; Test type: Superiority; p = 0.499, Fisher Exact; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.08 to 0.10]

7. Secondary Outcome: Number of Participants With Positive Cell Mediated Immune Response
Description: Cell mediated immune response was measured by interferon gamma (IFN-gamma) production by T-cells against each of the six HCV genotype 1b peptide pools in the vaccine. Positivity was defined as i) more than 48 spot forming cells per million PBMC; and ii) at least three times the mean background spots per million PBMC found in ELISpot wells containing cells and peptide diluent (DMSO). A participant was considered a responder if a positive response to at least one in 6 mixtures (pools) of peptides was detected.
Time Frame: Within 14 days after the last vaccination (Day 56)
Population: The population for this outcome included all participants who received both vaccinations and had immunogenicity data available. Participants are analyzed as treated. Data collected post-HCV infection were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
Number analyzed (Participants) | 125 | 122
Participants | 97 | 4

ADVERSE EVENTS:
Time Frame: Solicited reactogenicity symptoms were collected before vaccination, and then daily for 8 days post-vaccination (Day 0-7) after each vaccination on a memory aid. Unsolicited adverse events were collected through Day 90. At visits following Day 90 up to Day 140, only SAE's were collected.
Description: For events solicited on the memory aid, a participant was considered to have 1 event if it was reported as experienced at any time in the 8 day period after a vaccination. Participants are analyzed as treated, one participant randomized to placebo received vaccine.
Arm/Group | AdCh3NSmut1 and MVA-NSmut | Sodium Chloride Placebo
All-Cause Mortality (participants affected / at risk) | 5/274 | 2/272
Serious Adverse Events (participants affected / at risk) | 40/274 | 25/272
Other Adverse Events (participants affected / at risk) | 229/274 | 172/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdCh3NSmut1 and MVA-NSmut (N=274) | Sodium Chloride Placebo (N=272)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver Injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess Limb (Infections and infestations) | 2 (2) | 0 (0)
Abscess Neck (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bursitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
HIV Infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Psoas Abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foetal Monitoring (Investigations) | 1 (1) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Affective Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 3 (3) | 1 (1)
Schizoaffective Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 2 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdCh3NSmut1 and MVA-NSmut (N=274) | Sodium Chloride Placebo (N=272)
Injection site pain (General disorders) | 140 (176) | 21 (21) — Solicited as "Pain"
Injection site pain (General disorders) | 178 (247) | 43 (46) — Solicited as "Tenderness"
Injection site warmth (General disorders) | 52 (62) | 19 (21)
Injection site erythema (General disorders) | 95 (126) | 61 (77)
Injection site induration (General disorders) | 79 (98) | 29 (33)
Body temperature increase (Investigations) | 28 (29) | 8 (9)
Headache (Nervous system disorders) | 95 (114) | 64 (74)
Malaise (General disorders) | 114 (147) | 99 (120)
Myalgia (Musculoskeletal and connective tissue disorders) | 112 (138) | 69 (80)
Nausea (Gastrointestinal disorders) | 51 (64) | 48 (54)
Vomiting (Gastrointestinal disorders) | 26 (28) | 26 (29)
Chills (General disorders) | 51 (60) | 35 (40)
Abdominal pain (Gastrointestinal disorders) | 45 (57) | 34 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 (78) | 37 (45)
Aspartate aminotransferase increased (Investigations) | 29 (30) | 29 (31)
Blood alkaline phosphatase increased (Investigations) | 15 (15) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT01436357/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT01436357/SAP_001.pdf